CLINICAL TRIAL: NCT01412853
Title: Evaluation of the Response to Irradiation With MR-Spectroscopy for Localised Prostate Cancer Patients (The ERIS Trial)
Brief Title: Spectro-IRM and Evaluation Response to Prostatic Radiotherapy
Acronym: ERIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0203-1crgi 07/005-046
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: localized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (1):
- MR-spectroscopy (Experimental)
  Interventions: Other: MR-Spectroscopy

INTERVENTIONS:
Other: MR-Spectroscopy — response to standard radiotherapy treatment will be estimated for each patient every 3 months up to one year from the end of the radiotherapy

SUMMARY:
Context:

Prostate cancer is the most common non-cutaneous cancer and the second most common cause of cancer-related deaths in European and North-American men.

After external radiotherapy or brachytherapy, the Prostate Specific Antigen (PSA) value is often fluctuating and PSA nadir may only be reached after 2 years or more and may remain detectable several years after the completion of radiation. Moreover, PSA bounces and blips render patients and physicians very anxious about any possibility of a relapse. In this context, biomarkers that could predict the response to radiation earlier than PSA for patients with prostate cancer appear long overdue.

Magnetic Resonance Spectroscopy at 3 Tesla without endorectal coil is a non invasive procedure which allows quantification of metabolites such as Choline, Creatine, Polyamines and Citrate within the prostate gland.

Objectives:

The investigators are conducting a French prospective study on the Evaluation of the Response to Irradiation with MR Spectroscopy (ERIS). Their purpose is to monitor the early response of radiation with 3D MR Spectroscopy during the first year after completion of radiation and its impact on biochemical control. Therefore, the ERIS trial aims to investigate whether or not there could be a correlation between the time course of PSA and that of Choline and Citrate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a biopsy-proven prostatic adenocarcinoma
2. Gleason score between 4 and 10
3. Maximal baseline PSA < 50 ng/ml
4. Age over or = to 18 yr
5. Exclusive radiotherapy and/or brachytherapy with or without androgen deprivation therapy
6. Written informed consent from the patient

Exclusion Criteria:

1. lymph-node metastases
2. Bone metastases
3. Maximal baseline PSA ≥ 50 ng/ml
4. Prior radical prostatectomy
5. Contra-indications for MRI (Pace-maker, hip prothesis…)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
PSA value compare to Choline and Citrate levels as measured with MR-spectroscopic imaging as predictive factor of the response to treatment | up to 1 year
  Data will be collected at the end of the radiotherapy and every 3 months up to 1 year for each patient. Data analysis will be performed at the end of data completion in december 2011.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France